CLINICAL TRIAL: NCT00234988
Title: Safety and Weight Reduction of Sibutramine in the Treatment of Thai Obese and Overweight Subjects
Brief Title: A Phase IV, Multi-Center, Open-Label Trial of Sibutramine in Combination With a Hypocaloric Diet in Obese and Overweight Thai Subjects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, MD, PhD, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THAI-03-002
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Obesity
Keywords: Sibutramine; Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: sibutramine hydochloride monohydrate

INTERVENTIONS:
Drug: sibutramine hydochloride monohydrate — 10 mg QD with the option to increase dose to 15 mg QD up until Week 4
  Other Names: ABT-991; sibutramine; Meridia

SUMMARY:
The purpose of the study is to determine the safety and weight loss when sibutramine is used in overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has nutritional obesity and BMI >30 kg/m

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus
* Inadequately controlled hypertension
* History of Gilles de la Tourette's Syndrome.
* Use of any MAOIs, SSRIs, amino acids, antimigraine drugs, opioids
* Hypothyroidism or hyperthyroidism.
* History of:

  * benign prostatic hyperplasia
  * neurological disorders
  * psychiatric illness
  * severe renal or hepatic impairments
  * narrow-angle glaucoma
* History of cardiovascular disease or cerebrovascular disease
* Persistent tachycardia at rest
* Pulmonary hypertension
* Phaeochromocytoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2004-06; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 48 weeks
Safety parameters | 48 weeks

SECONDARY OUTCOMES:
Waist and hip circumference | 48 weeks
Fasting glucose | 48 weeks
Fasting lipids | 48 weeks
Uric acid | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 1-800-633-9110, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States